CLINICAL TRIAL: NCT04213495
Title: Czech Anesthesia Day 2019: Observational Trial
Brief Title: Czech Anesthesia Day 2019
Acronym: CAD2019
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Krajská zdravotní a.s. University Hospital Ústí nad Labem (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2019/12
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia Practice
Keywords: Anesthesia; Practice; Czech Republic
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing anesthesia in Czech Republic: Patients undergoing anesthesia in Czech Republic in the selected period from the confirmed Anesthesia Center
  Interventions: Other: Anesthesia

INTERVENTIONS:
Other: Anesthesia — Patients undergoing anesthesia from the cooperating Anesthesia center

SUMMARY:
Czech Anesthesia Day 2019 was designed as a prospective observational trial with the aim to evaluate the current anesthesiology practice in Czech Republic.

DETAILED DESCRIPTION:
Anesthesiology centers in Czech Republic was screened for cooperation during the year 2018. Data from centers with previously confirmed cooperation will be screened and filled into the electronic database. The basic information about the centre, patient´s demography, American Society of Anesthesiologist classification (ASA), type of surgery/anesthesia, airway management, type of anesthesia induction, drugs for anesthesia induction a and anesthesia maintenance, used monitors of vital signs and functions, type and amount of infusions, temperature management, intravenous lines management, patient blood management, mechanical ventilation settings and postoperative admission will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients from confirmed Anesthesiology Centers - previously confirmed the cooperation (center is registered in the online database with the unique identification)

Exclusion Criteria:

* Data from centers with not confirmed cooperation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical or diagnostic procedure under anesthesia in the Czech Republic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia description | From anesthesia induction until the admission to postanesthesia care
  Data from confirmed center will be recorded with the aim to describe the daily anesthesia practice in Czech Republic

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, assoc.Prof.MD.Ph.D, Study Chair — University Hospital Brno; Vladimir Cerny, Prof.MD.Ph.D., Study Director — Krajska zdravotni a.s. University Hospital Usti nad Labem
Locations (2):
- Czechia (2):
  - Brno University Hospital, Brno, South Moravian
  - Krajska zdravotni a.s. University Hospital Usti nad Labem, Ústí nad Labem

IPD SHARING:
Plan to Share IPD: Undecided